CLINICAL TRIAL: NCT02120976
Title: A Phase 1, Randomized, Single-blind, Placebo-controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) of Single Oral Doses of JTT-252 in Healthy Subjects (Part I); in Conjunction With an Open-label Study to Evaluate the Effect of Food on the PK of JTT-252 in Healthy Subjects (Part II); and an Open-label Study to Evaluate the Safety, Tolerability, PK and Pharmacodynamics (PD) of Single Oral Doses of JTT-252 in Type 2 Diabetic Subjects (Part III)
Brief Title: Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Doses of JTT-252
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT252-U-14-001
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus
Keywords: Safety; Tolerability; Pharmacokinetics; Food-effect; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (9):
- Dose 1 JTT-252 or Placebo (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252 or Placebo
- Dose 2 JTT-252 or Placebo (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252 or Placebo
- Dose 3 JTT-252 or Placebo (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252 or Placebo
- Dose 4 JTT-252 or Placebo (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252 or Placebo
- Dose 5 JTT-252 or Placebo (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252 or Placebo
- Dose 6 JTT-252 or Placebo (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252 or Placebo
- Dose 7 JTT-252 or Placebo (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252 or Placebo
- Dose 8 JTT-252 (Experimental): Tablets, single dose in fed condition
  Interventions: Drug: JTT-252
- Dose 9 JTT-252 (Experimental): Tablets, single dose in fasted condition
  Interventions: Drug: JTT-252

INTERVENTIONS:
Drug: JTT-252 or Placebo — Subjects will receive JTT-252 or Placebo
  Arms: Dose 1 JTT-252 or Placebo; Dose 2 JTT-252 or Placebo; Dose 3 JTT-252 or Placebo; Dose 4 JTT-252 or Placebo; Dose 5 JTT-252 or Placebo; Dose 6 JTT-252 or Placebo; Dose 7 JTT-252 or Placebo
Drug: JTT-252 — Subjects will receive JTT-252
  Arms: Dose 8 JTT-252; Dose 9 JTT-252

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK of single oral doses of JTT-252 and the effect of food on the PK of JTT-252 in healthy subjects, and to evaluate the safety, tolerability, PK and PD of single oral doses of JTT-252 in type 2 diabetes mellitus subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subject Cohorts:

* Healthy male or female subjects
* Age 18 to 50 Years (inclusive)
* Body Mass Index (BMI) between 19.0 and 31.0 kg/m2 (inclusive)

Type 2 Diabetic Subject Cohorts:

* Male or female Type 2 diabetic subjects who are currently being treated with a stable dose of metformin
* Age 18 to 65 Years (inclusive)
* BMI between 25.0 and 40.0 kg/m2 (inclusive)
* Have a glycosylated hemoglobin (HbA1c) of >7.0% to ≤9.5%
* Have a fasting plasma glucose (FPG) <240 mg/dL

Exclusion Criteria:

Healthy Subject Cohorts:

* Known clinically relevant history or presence of significant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, metabolic and dermatological or connective tissue disease
* Subjects with a systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg

Type 2 Diabetic Subject Cohorts:

* Subjects with a known medical history or presence of type 1 diabetes mellitus
* Subjects with known medical history of acute metabolic diabetic complications
* Subjects with uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >95 mmHg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 22 days
Vital signs and 12 lead ECGs | 22 days
Cmax (maximum concentration) | 22 days
t1/2 (elimination half-life) | 22 days
AUC (area under the concentration-time curve) | 22 days
fe(total) (fraction of systemically available drug excreted into the urine over entire collection interval) | 3 days
Plasma glucose | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Yuichiro Neki, Study Chair — Akros Pharma Inc.
Locations (2):
- United States (2):
  - Overland Park, Kansas
  - Austin, Texas